CLINICAL TRIAL: NCT06631222
Title: Effect of Cognitive Behaviour Approach on Subjects With Smartphone Addiction
Brief Title: to Stuidy the Effect of Cognitive Behavior Threapy CBT on Smartphone Addiction Patients With Tension Type Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hatem Mostafa (Other)
Responsible Party: Sponsor-Investigator, Hatem Mostafa, assistant lecturer of physical therapy, Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/120/005099
Record Dates: First submitted 2024-10-05; First posted 2024-10-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Tension Type Headache; Smartphone Addiction
MeSH Terms: conditions — Tension-Type Headache; Internet Addiction Disorder | interventions — Cognitive Behavioral Therapy; Manipulation, Spinal; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): the participants will receive a conventional standard physical therapy program (sub-occipital inhibitory pressure, Spinal manipulation, deep friction massage and corrective exercises)
  Interventions: Other: sub-occipital inhibitory pressure; Other: deep friction massage; Other: Spinal manipulation; Other: Exercises for forward head posture
- experimental group (Experimental): the participants will be treated with behavior change model in addition to a conventional standard physical therapy program for tension-type headache.
  Interventions: Behavioral: cognitive behavioral therapy; Other: sub-occipital inhibitory pressure; Other: deep friction massage; Other: Spinal manipulation; Other: Exercises for forward head posture

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — The therapeutic patient education (TPE) program was based on a biobehavioral approach and was divided into the following three parts: cognitive, operant, and respondent. The purpose of the TPE program was to modify erroneous beliefs about pain and disability, as well as to provide coping strategies and improve patient self-efficacy through a graded activity.
  Arms: experimental group
Other: sub-occipital inhibitory pressure — The suboccipital musculature will be palpated until contact is made with the posterior arch of the atlas, and progressive and deep gliding pressure was applied, pushing the atlas anteriorly. The occiput will be rested on the hands of the therapist while the atlas is supported by the fingertips. Finger pressure will be maintained for 10 minutes to produce the proposed therapeutic effect of inhibiting the suboccipital soft tissues.
Other: deep friction massage — Friction massage is performed with the fingertips placed on the trigger points. Pressure was applied and the fingertips move in a circular manner, while the pressure is gradually increased. This massage will be applied until the patient report a reduction in pain at the trigger point
Other: Spinal manipulation — This technique is performed along an imaginary vertical line passing through the odontoid process of the axis. No flexion or extension and very little lateral flexion will be used. Application will be bilateral. First, cephalic decompression will be performed lightly, followed by small circumductions. Selective tension will be applied to take up tissue slack and create a firm joint barrier. Manipulation is then performed with rotation towards the manipulated side in a helicoidal cranial movement. This technique will be applied with the aim of increasing occiput, atlas, and axis joint mobility.
Other: Exercises for forward head posture — Scapular stabilization exercises:
  1. In quadruped position, the patient lift¬ up his arms alternatively with shoulder abduction and 120 ° flexion.
  2. In sitting position, with 90° knee flexion on a stool or bed without backrest, patient hold a pair of dumb¬bells (2 kg) in each hand and lift them up laterally while maintaining scapulae's height below 80°. The patient was instructed to hold each stage for 10 seconds and then re-turn to the starting position and three sets of 10 repetitions with 30-second pause in between were completed.
  3. As for the progression of scapular stability exercise, T to Y the patient was instructed to lie in prone lying position on Swiss ball with arms abducted to 90° (the letter T); then she asked to flex elbows to 90°, retract scapulae and externally ro¬tate arms while keeping arm in 90° abductions. While maintaining the retraction of scapula, the patient is asked to raise his arms above head and extend the elbow while his arm flexed and abducted to 120°

SUMMARY:
The goal of this clinical trial is to learn if cognitive behavioral approach works to treat tension type headache in smartphone addiction in adults. The main questions it aims to answer are:

Is there an effect of adding cognitive behavior approach to physical therapy (manual therapy, corrective exercise therapy) on pain pressure threshold, forward head posture and headache intensity in smartphone addiction patients with tension-type headache? Researchers will compare adding cognitive behavior approach to physical therapy (manual therapy, corrective exercise therapy) to see if cognitive behavior approach works to treat tension type headache in smartphone addiction than physical therapy alone.

Participants will:

All participants will receive twelve treatment sessions (twice per week) in a 6 weeks period with a rest period of 48 to 72 hour between them.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were those diagnosed with tension type headache by neurologists based on the criteria of the International Headache Society.
* age between 19-34.
* International Headache Society diagnostic criteria of tension type headaches:
* Frequent ETTH or CTTH diagnosed, in both cases more than three months.
* Episodes of pain from 30 minutes to 7 days Fulfil 2 or more of the following characteristics:
* Bilateral location of pain.
* Non-pulsatile pain pressure.
* Pain mild to moderate.
* The headache does not increase with physical activity.
* The headache may be associated with pericranial tenderness.
* Controlled pharmacologically.
* Myofascial TrPs were bilaterally explored in upper trapezius, splenius capitis, sternocleidomastoid, masseter, superior oblique, levator scapulae and suboccipital muscles, TrP diagnosis was conducted following the diagnostic criteria:
* presence of a palpable taut band within a skeletal muscle.
* presence of a hypersensitive tender spot in the taut band.
* local twitch response elicited by snapping palpation of the taut band reproduction of the typical referred pain pattern of the TrP in response to compression.
* TrPs were considered active if both the local and the referred pain evoked by manual palpation reproduced total or partial pattern of the headache.
* Patients with FHP who have craniovertebral angle less than 49 degrees were included. Forward head posture is measured by calculating the angle between the horizontal line passing through C7 and a line extending from the tragus of the ear to C7.
* patients with smartphone addiction who will score 31 for males and 33 for females on smartphone addiction scale - short version.

Exclusion Criteria:

* rheumatoid arthritis.
* suspected malignancy.
* pregnancy.
* if they had received manual therapy treatment in the 2 months before enrolment into the study.
* Patients with infrequent episodic tension type headache, or with probable frequent and infrequent forms of tension type headache or other concomitant headache.
* They can never have vomiting or headache episodes during the treatment.
* Episodic tension type headache patients may experience very occasionally photophobia or phonophobia during their episodes of headache.
* Chronic tension type headache patients may experience very occasionally photophobia, phonophobia or mild nausea during headache episodes.
* Pain aggravated by movement of the head.
* Metabolic or musculoskeletal problems with similar headache symptoms.
* Previous trauma to the cervical spine.
* Active vertigo history.
* Poorly controlled hypertension.
* Atherosclerosis.
* Advanced osteoarthritis.
* Patients undergoing pharmacological adaptation or changes in the prophylactic medication.
* Excessive emotional stress.
* Patients with heart devices.
* Joint instability.
* Neurological disorders.
* Laxity of cervical soft tissues.
* Radiographic abnormalities.
* Generalized hyperlaxity or hypermobility.

Ages: 19 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
pressure algometer | from enrollment to nthe end of treatment at 6 weeks
  this device is used to describe the sensitivity of the trigger points found in cervical region

SECONDARY OUTCOMES:
measurement of forward head posture | from enrollment to nthe end of treatment at 6 weeks
  participants will be imaged at a distance of 1.5m from their sitting position, and the participant's shoulder and the camera height were placed at the same level. The CVA will be measured using a horizontal line passing through the C7 spinous process and a line connecting C7 to the tragus of the ear.
Headache impact test | from enrollment to nthe end of treatment at 6 weeks
  A popular patient-reported outcome measure for evaluating the detrimental effects of headaches on a patient's normal activity is the shortform Headache Impact Test. It was created before the FDA's now-accepted patient-reported guidance was established, utilizing the general headache population. HIT-6 was created for usage in a broad headache population and comprises of 6 elements. It gauges the frequency of recent headaches that were unbearably painful, interfered with everyday activities, made you want to lie down, or left you grouchy, exhausted, or unable to concentrate. higher values mean worse outcome while, lowered values menas better outcome
The smartphone addiction scale short version | from enrollment to nthe end of treatment at 6 weeks
  This scale is a short version that contains only 10 questions for easy smartphone addiction screening of adolescents who are considered vulnerable to addiction. This scale also provides a cut-off value to evaluate the level of addiction, to evaluate the treatment effect and to provide evidence of interventions different from those in the conventional scales. This scale has a high value as a screening tool because gender differences can be reflected in the results by providing a cut-off value for both genders, and the screening process that includes the evaluation by clinical psychologists is not merely the simple percentage calculation method but reflects the characteristics of the participants. The cut-off value for boys is 31, Meanwhile, the cut-off value, for girls is 33

CONTACTS AND LOCATIONS:
Locations (1):
- the British University in Egypt, Cairo, Cairo Governorate, Egypt